CLINICAL TRIAL: NCT04922138
Title: Efficacy and Safety of Aumolertinib as Adjuvant Therapy in Resectable Stage I NSCLC With High-grade Patterns and EGFR-sensitizing Mutations (APPOINT)
Brief Title: Aumolertinib Adjuvant Therapy of Resectable Stage I EGFRm+ NSCLC With High-grade Patterns
Acronym: APPOINT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baohui Han (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Baohui Han, Chief physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSM-10296-A017
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Orally 110 mg Aumolertinib tablets (55 mg/tablet, 2 tablets/day) once a day .
  Interventions: Drug: Aumolertinib
- Arm B (No Intervention): Observation

INTERVENTIONS:
Drug: Aumolertinib — All subjects who meet the enrollment conditions will be included in the Aumolertinib monotherapy group: Orally 110 mg Aumolertinib tablets (55 mg/tablet, 2 tablets/day) once a day until recurrence or completion of treatment or reaching the standard of discontinuation.
  Other Names: HS-10296
  Arms: Arm A

SUMMARY:
Efficacy and safety of postoperative adjuvant treatment of NSCLC patients with Aumolertinib.

DETAILED DESCRIPTION:
This is a multi-center, two-arm clinical study. In patients with stage I non-squamous non-small cell lung cancer (NSCLC) with EGFR 19del/21L858R with solid, micropapillary, and/or complex gland components ≥10% who have not received any systemic treatment, to evaluate the efficacy and safety of postoperative adjuvant Aumolertinib in NSCLC patients .

ELIGIBILITY:
Inclusion Criteria:

Any patient who meets all of the following inclusion criteria will qualify for entry into the study:

1. Male or female, aged at least 18 years.
2. Histologically confirmed diagnosis of primary non small lung cancer (NSCLC) on predominantly non-squamous histology.
3. Brain examination must be done prior to surgery as it is considered standard of care.
4. Patients are pathologically confirmed to be stage I after operation, containing solid, micropapillary, and/or complex gland components ≥10%.
5. Confirmation by the central laboratory that the tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including T790M.
6. Providing paraffin embedded section(10-15sheets),wax blocks or fresh frozen tissues.
7. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour.
8. World Health Organization Performance Status of 0 to 1.
9. Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after stopping the study treatment and should not breastfeed. Before starting the administration, the pregnancy test was negative.
10. Male patients should be willing to use barrier contraception from screening to stopping study treatment for 3 months.(i.e., condoms).
11. For inclusion in study, patient must provide a written informed consent.
12. ≤10 weeks between surgery and treatment period

Exclusion Criteria:

Any patient who meets any of the following exclusion criteria will not qualify for entry into the study:

1. Treatment with any of the following:

   1. Pre-operative or post-operative or planned radiation therapy for the current lung cancer
   2. Pre-operative (neo-adjuvant) platinum based or other chemotherapy
   3. Prior treatment with neoadjuvant or adjuvant EGFR-TKI at any time
   4. Any other anti-tumor treatment for lung cancer(Including proprietary Chinese patent medicine with anti-tumor effects and anti-tumor immunotherapy, etc.)
   5. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   6. Treatment with an investigational drug within five half-lives of the compound or any of its related material.
   7. Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug..
2. Patients who have had only segmentectomies or wedge resections
3. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years following the end of treatment.
4. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of Aumolertinib.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
8. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
9. Inadequate bone marrow reserve or organ function.
10. History of hypersensitivity to any active or inactive ingredient of Aumolertinib, or to drugs with a similar chemical structure or class to Aumolertinib.
11. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
12. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
2-year Disease free survival (DFS) rate | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Defined as the proportion of patients alive and disease free at 2 years,estimated from Kaplan Meier plots of the primary endpoint of DFS at the time of the primary analysis

SECONDARY OUTCOMES:
3-, 4-, and 5-year DFS rate | From date of treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Defined as the proportion of patients alive and disease free at 3, 4 and 5 years, respectively, estimated from Kaplan Meier plots of the primary endpoint of DFS at the time of the primary analysis.
Overall Survival (OS) | Start of study drug to Survival Endpoint through study completion, an average of 5 years, assessed up to 60 months
  Defined as the time from the date of treatment start until date of death due to any cause
Patient health-related quality of life and symptoms (HRQoL) by SF-36v2 Health Survey | From date of treatment start until treatment completion or discontinuation, assessed up to 60 months
  Defined as a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section and the scores range from 0-100. A score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) | From date of treatment start until 28 days after treatment completion
  AEs graded by CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No